CLINICAL TRIAL: NCT02078739
Title: Tele-Yoga for Chronic Obstructive Pulmonary Disease and Heart Failure Patients: A Pilot Study
Brief Title: Tele-yoga Program in COPD and Heart Failure
Acronym: Tele-yoga
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 12-08383; Tele-Yoga (Other Grant/Funding Number: UCSF School of Nursing)
Record Dates: First submitted 2014-02-24; First posted 2014-03-05 (Estimated); Last update posted 2015-01-27 (Estimated); Status verified 2015-01

CONDITIONS: Yoga; COPD; Congestive Heart Failure
Keywords: Yoga; COPD; Congestive Heart Failure
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Heart Failure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Yoga Program (Experimental): Yoga Program twice per week for 8 weeks
  Interventions: Behavioral: Yoga Program at home using internet technology
- Education (Active Comparator): Education once per week for 8 weeks
  Interventions: Behavioral: Yoga Program at home using internet technology

INTERVENTIONS:
Behavioral: Yoga Program at home using internet technology

SUMMARY:
The combined diagnosis of chronic obstructive pulmonary disease (COPD) and heart failure (HF) is common but often missed because of similarities in clinical presentation, risk factors, and patient characteristics. The concurrent presence of both diseases worsens the limitations in exercise capacity and quality of life that patients experience with either disease alone. This pilot study will test the feasibility of a yoga program conducted in patients' homes using multi-point interactive videoconferencing ("Tele- Yoga") for patients with combined COPD/HF diagnoses. The investigators hypothesize that patients who receive a yoga program at home, compared to an educational control group, will experience fewer physical symptoms and better quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patients with heart failure (HF) who also have COPD according to University of California San Francisco medical record documentation and would like to participate in a home yoga intervention and hospitalization within the past 24 months.
* Patients must: receive permission from their provider to participate in the study
* English-speaking
* Score of 3 on the Mini-Cog test
* Be between the ages of 40 and 85 years
* New York Heart Association Class I-III left ventricular systolic or diastolic HF
* Have moderate-severe COPD defined as post bronchodilator Forced Expiratory Volume (FEV1) in 1 sec < 80% predicted, FEV1/Forced Vital Capacity ratio < 70% and history of smoking
* TV, broadband internet connection, enough space to practice yoga in front of the TV, and willing to have research assistant install videoconferencing equipment.

Exclusion Criteria:

* Patients with a history of medication non-compliance as described by their provider
* Hospitalization within the last 3 months
* Myocardial infarction or recurrent angina within the last 6 months
* Severe stenotic valvular disease
* History of sudden cardiac death without subsequent automatic internal defibrillator placement
* Cognitive impairment
* Neuromuscular, orthopedic, or psychiatric illness that would interfere with yoga training
* Oxygen saturation <85% on 6 liters of nasal oxygen.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2013-06; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Feasibility of home yoga program as measured by the participants' perception of the quality of the broadband connection. | 8 weeks
  To evaluate the feasibility, acceptability, adherence rate of an 8-week, 1-hr biweekly Tele-Yoga intervention. Feasibility will be determined by the quality of the broadband connection, acceptability measured by participant satisfaction with the Yoga program and adherence measured by the number of times a participant participates in the yoga program.

SECONDARY OUTCOMES:
Physical Function | 8 weeks
  Estimate the effect of home-based Tele-Yoga on physical function (endurance, balance, strength, and activity) and symptoms (dyspnea, sleep, and fatigue) compared to attention control

CONTACTS AND LOCATIONS:
Overall Officials: Jill N Howie-Esquivel, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

REFERENCES:
- [Derived] Selman L, McDermott K, Donesky D, Citron T, Howie-Esquivel J. Appropriateness and acceptability of a Tele-Yoga intervention for people with heart failure and chronic obstructive pulmonary disease: qualitative findings from a controlled pilot study. BMC Complement Altern Med. 2015 Feb 7;15:21. doi: 10.1186/s12906-015-0540-8. PMID 25887324